CLINICAL TRIAL: NCT02033369
Title: Ventrostriatal Dopamine Release and Reward Motivation in MDD
Brief Title: Imaging Dopamine Release in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other); Research Foundation for Mental Hygiene, Inc. (Other); Mclean Hospital (Other); Icahn School of Medicine at Mount Sinai (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Franklin Schneier, Professor, New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: #6853; 1R01MH099322-01A1 (NIH)
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Results first posted 2017-11-21 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; MDD; depression; pramipexole
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Pramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pramipexole (Experimental): Six weeks of treatment with oral pramipexole, initiated at 0.25 mg/day and titrated to a maximum daily dose of 2.5 mg.
  Interventions: Drug: Pramipexole
- Healthy Control (No Intervention): Healthy volunteers were matched to MDD group subjects by age, gender, and ethnicity, and will have no lifetime psychiatric disorders.

INTERVENTIONS:
Drug: Pramipexole — Dose will be started at 0.125 mg bid, and increased by 0.25 mg/day every 3-4 days to a target range of 1.0 - 2.5 mg/day.
  Other Names: Mirapex (brand name)
  Arms: Pramipexole

SUMMARY:
This study aims to determine whether ventral striatal dopamine release is a mechanism of reward motivation in major depression, whether dopamine release is low in depression, and whether DA release and reward motivation predict response to dopamine-targeted treatment with pramipexole.

DETAILED DESCRIPTION:
Better understanding of the basic neurobiology of mood dysfunction appears necessary to enable further progress in the treatment of depression. Reward motivation (and the closely related construct of "reward learning") is a core neurobehavioral domain.(1,2) In major depressive disorder (MDD), low reward motivation is a key aspect of anhedonia, a cardinal symptom of MDD, and is related to resistance to treatment.(2,3) Although much has been learned about reward motivation's neurobiology and relevance to psychopathology, important gaps in our knowledge have impeded the application of basic science findings to improving treatment of MDD. Reward motivation in healthy subjects involves ventrostriatal (VST) dopamine (DA)(4,5), and reduced reward motivation is linked to MDD and anhedonia.(3,6) These data suggest that VST DA dysfunction might be present in MDD and manifested clinically by anhedonia. While DA neuroreceptor imaging studies have failed to verify this, they have been methodologically compromised. Limitations include imaging methods with poor resolution of functional striatal subregions, MDD samples heterogeneous for antidepressant use, and use of self-report measures of anhedonia, rather than objective behavioral testing of the specific domain of reward motivation. This will be the first study of both VST DA release (by PET imaging) and reward motivation, and will include patients with MDD and healthy volunteers. Reward motivation will be captured and operationalized as reward learning in a probabilistic reward task (prior to imaging). This will clarify if VST DA dysfunction is linked to impaired motivation in MDD. To test clinical implications in MDD patients, we will assess the relationship of VST DA release, reward motivation, and anhedonia to outcome of subsequent open label treatment with the DA D2 receptor agonist pramipexole.

ELIGIBILITY:
Inclusion Criteria:

* Weight between 44 kg and 115 kg
* Meets DSM-IV criteria for principal diagnosis of MDD, current major depressive episode, without psychotic features
* Score of >16 and <29 on 17-item Hamilton Rating Scale for Depression
* Psychotropic-naïve, as defined by lifetime <2 weeks treatment with antidepressants, anxiolytics or antipsychotics
* Able to tolerate a treatment-free period during study participation
* Able to provide informed consent

Exclusion Criteria:

* A principal diagnosis of any current Axis I psychiatric disorder other than the MDD
* Lifetime diagnosis of any psychotic disorder, bipolar disorder, mental retardation, attention deficit/hyperactivity disorder, or substance use disorders (including nicotine use disorders)
* Serious suicidal risk or history of violent behavior which would make participation in the protocol unsafe
* Any tobacco use in the prior three months (if not already excluded for abuse/dependence by #1)
* Illicit drug use in the prior three months, as evidenced by history or urine toxicology screen
* Women who are pregnant, nursing, postmenopausal, or using hormonal methods of birth control
* Women who are not using an effective birth control method or sexual abstinence during the ten days before the scan
* Any medical or neurological problem that might affect interpretation of findings or safety of participation (e.g., blood dyscrasias, lymphomas, hypersplenism, endocrinopathies, renal failure or chronic obstructive lung disease, malignancy, neurological diseases of the brain, history of seizures or head trauma), low hemoglobin (Hb < 12 gm/dL in males, Hb < 10.5 gm/dL in females))
* Blood donation within 4 weeks of study
* Metal implants or paramagnetic objects in the body that might affect safety of undergoing MRI (e.g., heart pacemaker, shrapnel, bullets, surgical prostheses or surgical clips), as determined in consultation with a neuroradiologist and according to the guidelines set forth in the reference: "Guide to MR procedures and metallic objects" Shellock; Lippincott Williams and Wilkins, NY, 2001
* More than one major risk factor for coronary artery disease (e.g. hyperlipidemia, sedentary lifestyle). Smokers are already excluded by #4 above, and diabetics by #8 above
* Systolic blood pressure > 140 or diastolic blood pressure > 90 based on at least two readings at rest
* History of untoward reaction to amphetamine or other stimulant medication, or pramipexole
* Any psychotropic treatment in the past 3 weeks (or depot medication in the past 6 months), except for lorazepam,which may be administered as needed prior to imaging day
* Current, past or anticipated exposure to radiation in the workplace, or participation in nuclear medicine procedures, including research protocols (In case of previous exposure to activity due to research studies, subjects will be eligible if all conditions listed below are fulfilled: 1) The injected dose and dosimetry of the radiotracer are known; 2) Except for research studies, the subject has not been exposed to radiation (workplace and medical); 3) Adding prior exposure to the exposure due to the study will result in a yearly cumulative exposure lower than the FDA limit for research studies
* Family history of schizophrenia in parents, siblings, or children
* Ongoing cognitive-behavioral or interpersonal psychotherapy for depression (Supportive therapy is not an exclusion)
* Ongoing treatment with cimetidine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Schneier, MD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanislow CA, Pine DS, Quinn KJ, Kozak MJ, Garvey MA, Heinssen RK, Wang PS, Cuthbert BN. Developing constructs for psychopathology research: research domain criteria. J Abnorm Psychol. 2010 Nov;119(4):631-9. doi: 10.1037/a0020909. PMID 20939653
- [Background] Treadway MT, Zald DH. Reconsidering anhedonia in depression: lessons from translational neuroscience. Neurosci Biobehav Rev. 2011 Jan;35(3):537-55. doi: 10.1016/j.neubiorev.2010.06.006. Epub 2010 Jul 11. PMID 20603146
- [Background] Vrieze E, Pizzagalli DA, Demyttenaere K, Hompes T, Sienaert P, de Boer P, Schmidt M, Claes S. Reduced reward learning predicts outcome in major depressive disorder. Biol Psychiatry. 2013 Apr 1;73(7):639-45. doi: 10.1016/j.biopsych.2012.10.014. Epub 2012 Dec 8. PMID 23228328
- [Background] Forbes EE, Hariri AR, Martin SL, Silk JS, Moyles DL, Fisher PM, Brown SM, Ryan ND, Birmaher B, Axelson DA, Dahl RE. Altered striatal activation predicting real-world positive affect in adolescent major depressive disorder. Am J Psychiatry. 2009 Jan;166(1):64-73. doi: 10.1176/appi.ajp.2008.07081336. Epub 2008 Dec 1. PMID 19047324
- [Background] Kumar P, Waiter G, Ahearn T, Milders M, Reid I, Steele JD. Abnormal temporal difference reward-learning signals in major depression. Brain. 2008 Aug;131(Pt 8):2084-93. doi: 10.1093/brain/awn136. Epub 2008 Jun 25. PMID 18579575
- [Background] Pizzagalli DA, Iosifescu D, Hallett LA, Ratner KG, Fava M. Reduced hedonic capacity in major depressive disorder: evidence from a probabilistic reward task. J Psychiatr Res. 2008 Nov;43(1):76-87. doi: 10.1016/j.jpsychires.2008.03.001. Epub 2008 Apr 22. PMID 18433774
- [Derived] Whitton AE, Reinen JM, Slifstein M, Ang YS, McGrath PJ, Iosifescu DV, Abi-Dargham A, Pizzagalli DA, Schneier FR. Baseline reward processing and ventrostriatal dopamine function are associated with pramipexole response in depression. Brain. 2020 Feb 1;143(2):701-710. doi: 10.1093/brain/awaa002. PMID 32040562
- [Derived] Schneier FR, Slifstein M, Whitton AE, Pizzagalli DA, Reinen J, McGrath PJ, Iosifescu DV, Abi-Dargham A. Dopamine Release in Antidepressant-Naive Major Depressive Disorder: A Multimodal [11C]-(+)-PHNO Positron Emission Tomography and Functional Magnetic Resonance Imaging Study. Biol Psychiatry. 2018 Oct 15;84(8):563-573. doi: 10.1016/j.biopsych.2018.05.014. Epub 2018 May 25. PMID 30041971

RESULTS

PARTICIPANT FLOW:
Groups:
- MDD Patients: Six weeks of treatment with oral pramipexole, initiated at 0.25 mg/day and titrated to a maximum daily dose of 2.5 mg.
  Pramipexole: Dose will be started at 0.125 mg bid, and increased by 0.25 mg/day every 3-4 days to a target range of 1.0 - 2.5 mg/day
- Healthy Controls: Individuals without depression
Period: Overall Study
Arm/Group | MDD Patients | Healthy Controls
Started | 26 | 26
Completed | 21 | 21
Not Completed | 5 | 5
Not completed — Physician Decision | 1 | 2
Not completed — Not a good demographic match | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline information was collected for 26 patients with MDD and 25 HC control subjects. One HC subject signed consent but was withdrawn from the study before completing any assessments due to not matching well.
Groups:
- Healthy Control Patients: Healthy control patients did not receive study medication and only have baseline measures.
- Total: Total of all reporting groups
Arm/Group | MDD Patients | Healthy Control Patients | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (6.1) | 26.5 (5.6) | 26.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13
Hamilton Rating Scale for Depression [Mean (Standard Deviation); unit: units on a scale] — Hamilton Rating Scale for Depression (HRSD), 17-item version. This standard scale will be used to assess severity of depression, looking at change in total score from baseline to week 6, rating severity of depression on a scale from 0 (least depression) to 50 (greatest depression)
  units on a scale | 20.3 (2.7) | 0.2 (0.4) | 10.4 (10.3)
Snaith Hamilton Pleasure Scale [Mean (Standard Deviation); unit: units on a scale] — Fourteen-item self-rated anhedonia scale. Items were comprised of statements that participants rated as "strongly disagree" (1), "disagree" (2), "agree" (3), or "strongly agree" (4). The lowest possible score was 14, the highest possible score was 56.
  units on a scale | 31.9 (6.5) | 18.9 (4.8) | 25.7 (8.7)
Temporal Experience of Pleasure Scale - Anticipatory Subscale [Mean (Standard Deviation); unit: units on a scale] — A validated self-rated subscale assessing anticipatory pleasure. It will be used for exploratory analyses of anhedonia.
  18 items were measured on a scale of 1 (very false for me) to 6 (very true for me). Higher scores indicate higher pleasure. Item scores were added for a lowest possible score of 18 and highest possible score of 108.
  units on a scale | 36.1 (8.0) | 49.0 (5.2) | 42.4 (9.3)
Mood and Anxiety Symptom Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Change in Mood and Anxiety Symptom Questionnaire, Short Form. A 62-item scale assessing anxiety and depression. Items were measured on a scale of 1-5, higher number indicating higher levels of symptoms.The lowest possible score was 62, and the highest 310.
  units on a scale | 174.5 (28.6) | 83.9 (13.3) | 130.1 (50.8)
Apathy Evaluation Rating Scale [Mean (Standard Deviation); unit: units on a scale] — A validated self-rated 18 item scale assessing apathy. Items were rated from 1 (not at all true) to 4 (very true). Higher scores indicate lower apathy, lower scores indicate higher apathy. Lowest possible score is 18, highest possible score is 72.
  units on a scale | 41.8 (9.7) | 23.8 (4.9) | 33.0 (11.8)
Clinical Global Impression Severity [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression - severity. Seven-point likert scale rating clinical severity of mental illness from 1 (least severe) to 7 ( most severe). Physician-rated scale. One item Population: Only 22 MDD patients started treatment. Healthy controls, as per study design, did not receive treatment.
  units on a scale | 3.9 (0.7) | 1.0 (0) | 1.9 (0.4)
Temporal Experience of Pleasure Scale - Consummatory Subscale [Mean (Standard Deviation); unit: units on a scale] — A validated self-rated subscale assessing consummatory pleasure. It will be used for exploratory analyses of anhedonia.
  18 items were measured on a scale of 1 (very false for me) to 6 (very true for me). Higher scores indicate higher pleasure. Item scores were added for a lowest possible score of 18 and highest possible score of 108.
  units on a scale | 29.9 (7.6) | 38.4 (7.2) | 34.1 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Rating Scale for Depression
Description: Hamilton Rating Scale for Depression (HRSD), 17-item version. This standard scale will be used to assess severity of depression, looking at change in total score from baseline to week 6, rating severity of depression on a scale from 0 (least depression) to 50 (greatest depression)
Time Frame: Baseline and 6 weeks
Population: Healthy control subjects were not assessed for outcome measures because by study design they received no therapeutic intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 22
units on a scale | 8.4 (5.4)

2. Secondary Outcome: Change in Snaith Hamilton Pleasure Scale
Description: Fourteen-item self-rated anhedonia scale. Items were comprised of statements that participants rated as "strongly disagree" (1), "disagree" (2), "agree" (3), or "strongly agree" (4). The lowest possible score was 14, the highest possible score was 56.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 22
units on a scale | 26 (7.51)

3. Secondary Outcome: Change in Temporal Experience of Pleasure Scale - Anticipatory Subscale
Description: A validated self-rated scale shown to assess anticipatory pleasure. It will be used for exploratory analyses of anhedonia.
  18 items were measured on a scale of 1 (very false for me) to 6 (very true for me). Higher scores indicate higher pleasure. Item scores were added for a lowest possible score of 18 and highest possible score of 108.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 22
units on a scale | 43.2 (7.9)

4. Secondary Outcome: Change in Mood and Anxiety Symptom Questionnaire, Short Form
Description: Change in Mood and Anxiety Symptom Questionnaire, Short Form. A 62-item scale assessing anxiety and depression. Items were measured on a scale of 1-5, higher number indicating higher levels of symptoms.The lowest possible score was 62, and the highest 310.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 22
units on a scale | 123.1 (36.3)

5. Secondary Outcome: Change in the Apathy Evaluation Rating Scale
Description: A validated self-rated 18 item scale assessing apathy. Items were rated from 1 (not at all true) to 4 (very true). Higher scores indicate lower apathy, lower scores indicate higher apathy. Lowest possible score is 18, highest possible score is 72.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 22
units on a scale | 31.7 (9.5)

6. Secondary Outcome: Change in Clinical Global Improvement - Severity Scale
Description: Seven-point Likert scale rating clinical severity of mental illness from 1 (least severe) to 7 ( most severe). Physician-rated scale. One item.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 22
units on a scale | 2.59 (1.10)

7. Secondary Outcome: Change in Temporal Experiences of Pleasure Scale -- Consummatory Subscale
Description: A validated self-rated scale shown to assess consummatory pleasure. It will be used for exploratory analyses of anhedonia.
  18 items were measured on a scale of 1 (very false for me) to 6 (very true for me). Higher scores indicate higher pleasure. Item scores were added for a lowest possible score of 18 and highest possible score of 108.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 22
units on a scale | 35.6 (6.6)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Information was collected on a side effect checklist, with each adverse event rated from 0 (absent) to 3 (severe). A subject was considered to have experienced a side effect during the study if the rating for that adverse event increased in severity at any point during the treatment.
  Adverse events were not assessed for Healthy Controls, because by study design they did not receive any therapeutic intervention.
Groups:
- MDD Patients: Only patients with MDD received treatment. There was only one arm.
Arm/Group | MDD Patients
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDD Patients (N=22)
headache (Nervous system disorders) | 13 (13)
nausea (Gastrointestinal disorders) | 18 (18)
Heartburn (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 7 (7)
Decreased Appetite (Gastrointestinal disorders) | 6 (6)
Increased Appetite (Gastrointestinal disorders) | 6 (6)
Dry Mouth (General disorders) | 10 (10)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Sweating (Skin and subcutaneous tissue disorders) | 4 (4)
Skin Problems (Skin and subcutaneous tissue disorders) | 5 (5)
Bruising (Blood and lymphatic system disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 9 (9)
tremor (Musculoskeletal and connective tissue disorders) | 2 (2)
Impaired Coordination (Musculoskeletal and connective tissue disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 9 (9)
fatigue (General disorders) | 2 (2)
somnolence (Psychiatric disorders) | 11 (11)
Sleep Attacks (Psychiatric disorders) | 5 (5)
decreased libido (Reproductive system and breast disorders) | 7 (7)
Sexual Dysfunction (Reproductive system and breast disorders) | 3 (3)
Blurry Vision (Eye disorders) | 6 (6)
Lightheadedness (Nervous system disorders) | 10 (10)
Dizziness (Nervous system disorders) | 8 (8)
Forgetfulness (Psychiatric disorders) | 7 (7)
Impaired Concentration (Psychiatric disorders) | 2 (2)
compulsive behaviorws (Psychiatric disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No